CLINICAL TRIAL: NCT01792388
Title: Vitamin D and Its Effects on Inflammation and Intestinal Permeability in Crohn's Disease in Remission
Brief Title: Vitd and Barrier Function in IBD
Acronym: VIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: University of Calgary (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Tara Raftery, Dr. Maria O'Sullivan, PhD, University of Dublin, Trinity College
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: vip
Record Dates: First submitted 2012-12-19; First posted 2013-02-15 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Vitamin D; Intestinal Permeability; Tara Raftery
MeSH Terms: conditions — Crohn Disease | interventions — Vitamin D; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soya Bean oil (Placebo Comparator)
  Interventions: Dietary Supplement: Soya Bean oil
- Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Capsule Form
  Arms: Vitamin D
Dietary Supplement: Soya Bean oil — Capsule form
  Arms: Soya Bean oil

SUMMARY:
Increased Intestinal Permeability is detectable in clinically active Crohn's disease, in stable Crohn's disease and is predictive of clinical relapse. Maintenance of the epithelial barrier integrity is therefore essential for intestinal homeostasis. Vitamin D may have a critical role in improving barrier function.

ELIGIBILITY:
Inclusion Criteria:

* All patients must fulfill the clinical criteria for diagnosis of CD as defined by Lennard-Jones et al. (1976)
* All patients must be in clinical remission for at least 1 month at study entry as defined by a Crohn's Disease Activity Index (CDAI) of <150
* 18-65 years
* Patients on stable drug therapies for at least 1 month pre-enrolment
* Sufficient English language ability to carry out the study requirements

Exclusion Criteria:

* Symptomatic CD at study entry including CDAI >150
* Pregnancy
* Previous extensive small bowel resection (less than 200 cm of viable small bowel or a loss of 50% or more of the small intestine)
* Presence of an ileostomy or colostomy
* Known hypersensitivity to vitamin D
* Hypercalcaemia (corrected serum calcium > 2.66 mmol/L)
* Those currently using supplemental vitamin D >800 IU/D
* Diagnosis of any of the following: active tuberculosis, sarcoidosis, hyperparathyroidism, renal failure, pseudohyperparathyroidism, malignancy, active, lymphoma, short bowel syndrome
* Antibiotic use in the 4 weeks prior to enrolment
* Current use of bisphosphonates
* Renal Impairment, Diabetes Mellitus
* Patients participating in a concurrent RCT
* Alcohol dependency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Intestinal Permability from baseline and 3 months | 0 and 3 months
  Lactulose, Mannitol, Sucralose Test

SECONDARY OUTCOMES:
Change in Inflammatory and antimicrobial peptide levels from baseline to 3 months | Baseline and 3months
To assess change in grip strength and associated fatigue markers | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria O'Sullivan, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (2):
- Ireland (2):
  - Adelaide and Meath Hospital, Dublin
  - Tallaght Hospital, Dublin

REFERENCES:
- [Derived] Raftery T, Martineau AR, Greiller CL, Ghosh S, McNamara D, Bennett K, Meddings J, O'Sullivan M. Effects of vitamin D supplementation on intestinal permeability, cathelicidin and disease markers in Crohn's disease: Results from a randomised double-blind placebo-controlled study. United European Gastroenterol J. 2015 Jun;3(3):294-302. doi: 10.1177/2050640615572176. PMID 26137304